CLINICAL TRIAL: NCT02126670
Title: ACT01 in Combination With Comp01-04 in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP1401
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Investigator

ARMS (4):
- ACT01 plus Comp01 (Placebo Comparator): ACT01 Cream in combination with Comp01 Cream, once daily, 29 days
  Interventions: Drug: ACT01; Drug: Comp01
- ACT01 plus Comp02 (Active Comparator): ACT01 Cream in combination with Comp02 Cream, once daily, 29 days
  Interventions: Drug: ACT01; Drug: Comp02
- ACT01 plus Comp03 (Active Comparator): ACT01 Cream in combination with Comp03 Cream, once daily, 29 days
  Interventions: Drug: ACT01; Drug: Comp03
- ACT01 plus Comp04 (Other): ACT01 Cream in combination with Comp04 Cream, once daily, 29 days
  Interventions: Drug: ACT01; Drug: Comp04

INTERVENTIONS:
Drug: ACT01
Drug: Comp01
  Arms: ACT01 plus Comp01
Drug: Comp02
  Arms: ACT01 plus Comp02
Drug: Comp03
  Arms: ACT01 plus Comp03
Drug: Comp04
  Arms: ACT01 plus Comp04

SUMMARY:
The purpose of this study is to determine whether or not ACT01 is effective and tolerable alone or when used in combination with Comp01, Comp02, Comp03 or Comp04 in patients with facial and/or scalp keratosis.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of actinic keratosis lesions on the face and/or scalp within a 25 cm2 contiguous area containing at least four lesions that are non-hypertrophic and non-hyperkeratotic and not larger than 6 mm in longest diameter.
2. Age 30-85 years, inclusive.
3. Good general health as determined by investigator and supported by medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Severe, uncontrolled auto-immune, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, pulmonary or renal disease.
2. Dermatologic conditions if present on the face such as acne, atopic dermatitis, seborrheic dermatitis, eczema, rosacea, or albinism.
3. Application of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) UVB therapy to the intended treatment area within 180 days prior to the Baseline Visit.
4. Use of sun lamps or sun tanning beds or booths during the 14 days prior to the Baseline Visit.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Therapeutics Clinical Research, San Diego, California
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - Dermatology Consulting Services; Zoe Diana Draelos, MD, High Point, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- ACT01 Plus Comp01: ACT01 Cream in combination with Comp01 Cream, once daily, 29 days
  ACT01
  Comp01
- ACT01 Plus Comp02: ACT01 Cream in combination with Comp02 Cream, once daily, 29 days
  ACT01
  Comp02
- ACT01 Plus Comp03: ACT01 Cream in combination with Comp03 Cream, once daily, 29 days
  ACT01
  Comp03
- ACT01 Plus Comp04: ACT01 Cream in combination with Comp04 Cream, once daily, 29 days
  ACT01
  Comp04
Period: Overall Study
Arm/Group | ACT01 Plus Comp01 | ACT01 Plus Comp02 | ACT01 Plus Comp03 | ACT01 Plus Comp04
Started | 26 | 24 | 25 | 25
Completed | 25 | 24 | 25 | 24
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT01 Plus Comp01 | ACT01 Plus Comp02 | ACT01 Plus Comp03 | ACT01 Plus Comp04 | Total
Number analyzed (Participants) | 25 | 24 | 25 | 24 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.08) | 64.4 (9.78) | 66.5 (8.94) | 66.9 (8.28) | 65.5 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 7 | 2 | 18
  Male | 19 | 21 | 18 | 22 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 24 | 25 | 23 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 25 | 24 | 24 | 24 | 97
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 25 | 24 | 98

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success at End of Study Visit
Description: Treatment success at end of study visit defined as % of participants with 100% clearance of AK lesions
Time Frame: up to Day 57
Population: Per protocol
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACT01 Plus Comp01 | ACT01 Plus Comp02 | ACT01 Plus Comp03 | ACT01 Plus Comp04
Number analyzed (Participants) | 24 | 23 | 25 | 24
percentage of participants | 66.7 [47.8 to 85.5] | 65.2 [45.8 to 84.7] | 76.0 [59.3 to 92.7] | 66.7 [47.8 to 85.5]
Statistical Analysis 1: Comparison: ACT01 Plus Comp01 vs ACT01 Plus Comp02 vs ACT01 Plus Comp03 vs ACT01 Plus Comp04; Test type: Superiority or Other; p = 0.799, Chi-squared

2. Secondary Outcome: Irritation Score
Description: Percentage of participants with moderate or severe overall irritation at end of treatment.
Time Frame: up to Day 57
Population: Overall irritation
Measure: Number; unit: percentage of participants
Arm/Group | ACT01 Plus Comp01 | ACT01 Plus Comp02 | ACT01 Plus Comp03 | ACT01 Plus Comp04
Number analyzed (Participants) | 25 | 24 | 25 | 24
percentage of participants | 56.0 | 75.0 | 52.0 | 66.7

ADVERSE EVENTS:
Arm/Group | ACT01 Plus Comp01 | ACT01 Plus Comp02 | ACT01 Plus Comp03 | ACT01 Plus Comp04
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 22/26 | 24/24 | 20/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT01 Plus Comp01 (N=26) | ACT01 Plus Comp02 (N=24) | ACT01 Plus Comp03 (N=25) | ACT01 Plus Comp04 (N=25)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT01 Plus Comp01 (N=26) | ACT01 Plus Comp02 (N=24) | ACT01 Plus Comp03 (N=25) | ACT01 Plus Comp04 (N=25)
Application Site Irritation (General disorders) | 22 (22) | 24 (24) | 20 (20) | 24 (24)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No